CLINICAL TRIAL: NCT02208206
Title: Neuropathic Pain: Association Between Phenotype and Biomarkers
Brief Title: Analysis of Markers in the Blood Correlated With Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Christoph Stein, MD (Other)
Collaborators: deCODE genetics (Industry)
Responsible Party: Sponsor-Investigator, Christoph Stein, MD, Clinical director, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: NeuroPain CBF_01
Record Dates: First submitted 2014-07-29; First posted 2014-08-04 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Neuropathy
Keywords: Neuropathic pain; Phenotype; Genotype; Biomarkers; HIV; Diabetes mellitus; Breast cancer; Genomics; Quantitative sensory testing
MeSH Terms: conditions — Neuralgia; Diabetes Mellitus; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to analyze associations between symptoms and specific markers in the blood in patients suffering from neuropathic pain linked to diseases of different origin. Such markers could be utilized in the future for precise diagnosis of neuropathic pain and might lead to targeted pain treatment.

DETAILED DESCRIPTION:
On average, 3-8% of the German population suffers from neuropathic pain, which can occur after damage of somatosensory nerves in the peripheral or central nervous system. In terms of a "personalized" medicine, only a strict separation of neuropathic and chronic pain allows an individualized therapy to reduce pain severity and to enhance patients' quality of life.

Currently, the diagnosis of neuropathic pain is based on the medical history, the subjective description of somatosensory symptoms and the application of (non-genetic) diagnostic tests. To improve diagnosis and therapy of complex disorders for individual patients, novel methods are introduced based on flow cytometric (FACS) analysis of human immune cells or analysis of the human genome (genomics). Those techniques can support the identification of characteristic features indicating ongoing individual pathophysiologic processes in the body (biomarkers).

Often diseases are based on a complex relationship between genetics, environmental factors and the manifestation of the disease. To capture this complexity via genomics, phenotypical and genotypical data of high quality and detailed information about the study population are required.

This observational study includes patients suffering from painful and non-painful neuropathies associated with HIV-infection, diabetes mellitus and breast cancer. With the targeted application of validated questionnaires (such as the Brief Pain Inventory, Pain Catastrophizing Scale, Hospital Anxiety and Depression Scale, Ten-Item Personality Inventory, 36-Item Short Form Health Survey, and the Insomnia Severity Index) and parallel usage of genomics or FACS analysis of selected biomarkers in the blood, this study will provide information about the manifestation of certain genes or immune markers which are directly correlated to the symptoms of the disease. Additional performance of neuropsychological/cognitive tests and quantitative sensory testing (QST) will enhance the phenotypic profile. Identification of potential indicators could be utilized prospectively to precisely diagnose and effectively treat neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* HIV-associated neuropathy
* Sufficient knowledge of the German language

Exclusion Criteria:

* Co-incident severe central nervous system diseases
* Major psychiatric conditions
* Dementia
* Limited mental capacity or limited German language skills
* Intoxication with alcohol or recreational drugs within the last 48 hours of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals, primary care clinics, resident physicians
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Analysis of gene expression | Assessment - 1 day
  Investigation of associations between phenotypic and genotypic data. Patients with chronic painful and non-painful neuropathy will be phenotyped in detail using validated questionnaires related to pain (Brief Pain Inventory and Numeric Rating Scale), mental health (Pain Catastrophizing Scale and Hospital Anxiety and Depression Rating Scale), personality (Ten-Item Personality Inventory) and quality of life (36-Item Short Form Health Survey and Insomnia Severity Index). Optional, a set of neuropsychological/cognitive tests and quantitative sensory testing (QST) will be performed. DNA will be isolated from patients' blood samples and analyzed for genetic variants which might have an effect on the development of neuropathic pain. Once, phenotypic and genotypic data are available they will be associated with each other with the goal to find genetic variants tied to pain phenotypes and which might serve as novel DNA biomarkers for neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stein, Prof., Principal Investigator — Department of Anesthesiology Charite
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine, Charité - Universitätsmedizin Berlin, Berlin, Germany